CLINICAL TRIAL: NCT03649399
Title: Sonographic Detection of Pancreatic Stents Placed for Prophylaxis of Post-ERCP Pancreatitis
Brief Title: Sonographic Detection of Prophylactic Pancreatic Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, Prof., Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 419/17
Record Dates: First submitted 2018-08-25; First posted 2018-08-28 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pancreatitis; Stent Dislodgement
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pancreatic stent (Experimental): abdominal ultrasound and x-ray for stent detection.
  Interventions: Diagnostic Test: Abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Abdominal ultrasound — Abdominal ultrasound for detection of the pancreatic stent

SUMMARY:
The Retention of pancreatic stents for prophylaxis of post-ERCP pancreatitis (PEP) is assessed by abdominal x-ray according to international Guidelines. The current study aimed to analyze whether prophylactic pancreatic stents can be detected by transdermal ultrasound to save the x-ray examination.

DETAILED DESCRIPTION:
Pancreatitis is the most common complication of endoscopic retrograde cholangiopancreatography (ERCP). Several pharmacologic and procedure-related measurements have been established for post-ERCP pancreatitis (PEP) prophylaxis one being the placement of pancreatic duct stents in patients with high risk for PEP. The beneficial role of pancreatic stenting in the prophylaxis of PEP was demonstrated in large meta-analyses. The used stents have a high potential of self dislodgment, retained stents have to be removed endoscopically after 5-10 days. For evaluation of spontaneous stent passage abdominal x-ray ist used and accordingly retained stents removed. The current study aimed to analyze whether prophylactic pancreatic stents can be detected by transdermal ultrasound to save the x-ray examination.

ELIGIBILITY:
Inclusion Criteria:

* patient after pancreatic stent placement for prophylaxis of post-ERCP pancreatitis
* age 18-79
* signed informed consent

Exclusion Criteria:

* any disease that rules out study participation
* patient not legally competent to sign informed consent
* chronic pancreatis as indication for pancreatic stenting

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of the sonographic detection of pancreatic stents | 5-10 days after stent placement
  Test whether the stents can be detected reliably by ultrasound

SECONDARY OUTCOMES:
Negative predictive value of the sonographic detection of pancreatic stents | 5-10 days after stent placement
  Test whether and why the stents cannot be detected reliably by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, MD, Principal Investigator — Goethe University
Locations (1):
- Klinikum der J.W. Goethe-Universität, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michael FA, Gerber L, Weiler N, Hunyady PM, Abedin N, de la Vera AL, Stoffers P, Filmann N, Zeuzem S, Bojunga J, Friedrich-Rust M, Dultz G. Transabdominal ultrasonography to reduce the burden of X-ray imaging in prophylactic pancreatic stent localization after ERCP-A prospective trial. United European Gastroenterol J. 2021 May;9(4):469-477. doi: 10.1002/ueg2.12063. Epub 2021 Apr 22. PMID 33887119